CLINICAL TRIAL: NCT05270720
Title: Dendritic Cell Vaccination for the Adult Ovarian Cancer
Brief Title: Dendritic Cell Vaccination With Standard Postoperative Chemotherapy for the Treatment of Adult Ovarian Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: West China Second University Hospital (Other)
Responsible Party: Principal Investigator, Rutie Yin, Clinical Professor, West China Second University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WCSUH2022001
Record Dates: First submitted 2022-02-12; First posted 2022-03-08 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-02

CONDITIONS: Recurrent Ovarian Cancer
Keywords: neoantigen; dendritic cell vaccine
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental group (Experimental): This arm will evaluate the safety of administering a total dendritic cell dose of 5x106. A total of 3 to 6 patients will be enrolled. If this dose is associated with unacceptable side effects, as detailed in the study protocol, no further patients will be enrolled at this dose.
  Interventions: Biological: dendritic cell

INTERVENTIONS:
Biological: dendritic cell — Biological: Dendritic Cell Immunotherapy Adult patients with histopathologically diagnosed Ovarian Cancer will be eligible for this novel, personalized dendritic cell vaccine during course of standard of care chemotherapy.
  If unacceptable side effects are observed at a total dose of 5x106, as detailed in the study protocol, then a cohort of 3-6 enrolled patients will receive a de-escalated total dendritic cell dose of 2.5x106.
  If no unacceptable side effects are identified at a total dose of 5x106, as detailed in the study protocol, then a cohort of 3-6 enrolled patients will receive an escalated total dendritic cell dose of 1X107.

SUMMARY:
Effective treatments are desperately needed for ovarian cancer patients. This phase I clinical trial assesses the safety of a novel personalized dendritic-cell vaccine administered to ovarian cancer patients. Secondary outcomes will be evaluated such as patient pharmacodynamics， progression-free survival and overall survival.

DETAILED DESCRIPTION:
This is a single arm, non-randomized phase I study to evaluate the safety and feasibility of delivering a novel dendritic cell vaccine in 6 to 12 (n=6-12) adult patients diagnosed with ovarian cancer after undergoing surgical resection. The vaccine contains both tumor-associated antigen and patient specific neoantigens. Standard-of-care chemotherapy therapy will be followed as per routine,during which patients enrolled into this study will receive a personalized vaccine in addition to standard of care. Effective adjuvant therapies are urgently needed for these patients given that high rate of recurrence still occurs after standard of care with poor prognosis among ovarian cancer patients. The study is constructed in a 3+3 algorithm for two steps of dose escalation with rigorous and mandatory safety monitoring.

ELIGIBILITY:
Inclusion Criteria:

1. 18-75 years old female patients；
2. Histopathologically diagnosed recurrent stage III/IV epithelial ovarian cancer;
3. Normal liver, heart as well as kidney functions and blood chemistry;
4. Predicted survival for more than 6 months；
5. Provision of signed and dated informed consent form.

Exclusion Criteria:

1. Allergic to human albumin, an excipient of the manufactured dendric cell vaccine；
2. Predicted survival for less than 6 months；
3. Diagnosed with brain metastasis and other diseases unsuitable for cell therapy including but not limited to Myelodysplastic Syndromes、Acute Myeloid Leukemia and Systemic Lupus Erythematosus;
4. Diagnosed with viral diseases including but not limited to HIV, TP, HCV and HBV ；
5. Female patients who are pregnant, breast feeding, or of childbearing potential without a negative pregnancy test prior to baseline;
6. Other conditions deemed unsuitable for this study by the leading investigators.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 9 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
adverse events | up to 18 months
  Patients will be monitored for adverse events as dictated by CTCAE version 5.

SECONDARY OUTCOMES:
Pharmacodynamics | up to 1 week
  percentage of antigen-specific T cells in peripheral blood.
PFS | up to 18 months
  Progression-free survival
OS | up to 18 months
  Overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- west china second University， SICHUAN University, China, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anguille S, Van de Velde AL, Smits EL, Van Tendeloo VF, Juliusson G, Cools N, Nijs G, Stein B, Lion E, Van Driessche A, Vandenbosch I, Verlinden A, Gadisseur AP, Schroyens WA, Muylle L, Vermeulen K, Maes MB, Deiteren K, Malfait R, Gostick E, Lammens M, Couttenye MM, Jorens P, Goossens H, Price DA, Ladell K, Oka Y, Fujiki F, Oji Y, Sugiyama H, Berneman ZN. Dendritic cell vaccination as postremission treatment to prevent or delay relapse in acute myeloid leukemia. Blood. 2017 Oct 12;130(15):1713-1721. doi: 10.1182/blood-2017-04-780155. Epub 2017 Aug 22. PMID 28830889
- [Background] Carreno BM, Magrini V, Becker-Hapak M, Kaabinejadian S, Hundal J, Petti AA, Ly A, Lie WR, Hildebrand WH, Mardis ER, Linette GP. Cancer immunotherapy. A dendritic cell vaccine increases the breadth and diversity of melanoma neoantigen-specific T cells. Science. 2015 May 15;348(6236):803-8. doi: 10.1126/science.aaa3828. Epub 2015 Apr 2. PMID 25837513
- [Background] Liau LM, Ashkan K, Tran DD, Campian JL, Trusheim JE, Cobbs CS, Heth JA, Salacz M, Taylor S, D'Andre SD, Iwamoto FM, Dropcho EJ, Moshel YA, Walter KA, Pillainayagam CP, Aiken R, Chaudhary R, Goldlust SA, Bota DA, Duic P, Grewal J, Elinzano H, Toms SA, Lillehei KO, Mikkelsen T, Walbert T, Abram SR, Brenner AJ, Brem S, Ewend MG, Khagi S, Portnow J, Kim LJ, Loudon WG, Thompson RC, Avigan DE, Fink KL, Geoffroy FJ, Lindhorst S, Lutzky J, Sloan AE, Schackert G, Krex D, Meisel HJ, Wu J, Davis RP, Duma C, Etame AB, Mathieu D, Kesari S, Piccioni D, Westphal M, Baskin DS, New PZ, Lacroix M, May SA, Pluard TJ, Tse V, Green RM, Villano JL, Pearlman M, Petrecca K, Schulder M, Taylor LP, Maida AE, Prins RM, Cloughesy TF, Mulholland P, Bosch ML. First results on survival from a large Phase 3 clinical trial of an autologous dendritic cell vaccine in newly diagnosed glioblastoma. J Transl Med. 2018 May 29;16(1):142. doi: 10.1186/s12967-018-1507-6. PMID 29843811
- [Background] Ott PA, Hu-Lieskovan S, Chmielowski B, Govindan R, Naing A, Bhardwaj N, Margolin K, Awad MM, Hellmann MD, Lin JJ, Friedlander T, Bushway ME, Balogh KN, Sciuto TE, Kohler V, Turnbull SJ, Besada R, Curran RR, Trapp B, Scherer J, Poran A, Harjanto D, Barthelme D, Ting YS, Dong JZ, Ware Y, Huang Y, Huang Z, Wanamaker A, Cleary LD, Moles MA, Manson K, Greshock J, Khondker ZS, Fritsch E, Rooney MS, DeMario M, Gaynor RB, Srinivasan L. A Phase Ib Trial of Personalized Neoantigen Therapy Plus Anti-PD-1 in Patients with Advanced Melanoma, Non-small Cell Lung Cancer, or Bladder Cancer. Cell. 2020 Oct 15;183(2):347-362.e24. doi: 10.1016/j.cell.2020.08.053. PMID 33064988
- [Result] Harari A, Graciotti M, Bassani-Sternberg M, Kandalaft LE. Antitumour dendritic cell vaccination in a priming and boosting approach. Nat Rev Drug Discov. 2020 Sep;19(9):635-652. doi: 10.1038/s41573-020-0074-8. Epub 2020 Aug 6. PMID 32764681
- [Result] Zhang W, Lu X, Cui P, Piao C, Xiao M, Liu X, Wang Y, Wu X, Liu J, Yang L. Phase I/II clinical trial of a Wilms' tumor 1-targeted dendritic cell vaccination-based immunotherapy in patients with advanced cancer. Cancer Immunol Immunother. 2019 Jan;68(1):121-130. doi: 10.1007/s00262-018-2257-2. Epub 2018 Oct 10. PMID 30306202
- [Result] Tanyi JL, Bobisse S, Ophir E, Tuyaerts S, Roberti A, Genolet R, Baumgartner P, Stevenson BJ, Iseli C, Dangaj D, Czerniecki B, Semilietof A, Racle J, Michel A, Xenarios I, Chiang C, Monos DS, Torigian DA, Nisenbaum HL, Michielin O, June CH, Levine BL, Powell DJ Jr, Gfeller D, Mick R, Dafni U, Zoete V, Harari A, Coukos G, Kandalaft LE. Personalized cancer vaccine effectively mobilizes antitumor T cell immunity in ovarian cancer. Sci Transl Med. 2018 Apr 11;10(436):eaao5931. doi: 10.1126/scitranslmed.aao5931. PMID 29643231
- [Derived] Wang W, Jiang J, Yang C, Meng X, Gao L, Yuan Y, Lei T, Ding P, Yin R, Li Q. A critical time window for leukapheresis product transportation to manufacture clinical-grade dendritic cells with optimal anti-tumor activities. Cytotherapy. 2024 Feb;26(2):210-220. doi: 10.1016/j.jcyt.2023.12.003. Epub 2023 Dec 19. PMID 38127032
- [Derived] Li Q, Yang C, Tian H, Jiang J, Li P, Zhu X, Lei T, Yin R, Ding P, Bai P, Li Q. Development of a personalized dendritic cell vaccine and single-cell RNA sequencing-guided assessment of its cell type composition. Cytotherapy. 2023 Feb;25(2):210-219. doi: 10.1016/j.jcyt.2022.10.013. Epub 2022 Nov 25. PMID 36443171